CLINICAL TRIAL: NCT06222268
Title: Wayne State Warriors Marijuana Clinical Research Program: Cannabinoid Adjunct to Prolonged Exposure & Recovery
Acronym: CAPER
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Christine Rabinak, PhD, Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB-23-05-5773
Record Dates: First submitted 2023-10-13; First posted 2024-01-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: PTSD; Post Traumatic Stress Disorder
Keywords: Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cannabidiol; Single Person; nabiximols; Sugars; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (PBO) only (Placebo Comparator): In a double-blind, placebo and active-controlled, between-subjects design, the investigators will administer drugs containing THC (2.5mg), CBD (2.5mg) or PBO (0mg THC/CBD). Drug is administered and smoked immediately prior to exposure therapy sessions 3-6. 70 participants will be randomly assigned to each treatment arm. All participants will receive prolonged exposure therapy.
  Interventions: Drug: Placebo only
- Cannabidiol (CBD) only (Experimental): In a double-blind, placebo and active-controlled, between-subjects design, the investigators will administer drugs containing THC (2.5mg), CBD (2.5mg) or PBO (0mg THC/CBD). Drug is administered and smoked immediately prior to exposure therapy sessions 3-6. 70 participants will be randomly assigned to each treatment arm. All participants will receive prolonged exposure therapy.
  Interventions: Drug: Cannabidiol (CBD) only
- Delta-9-tetrahydrocannabinol (THC) only (Experimental): In a double-blind, placebo and active-controlled, between-subjects design, the investigators will administer drugs containing THC (2.5mg), CBD (2.5mg) or PBO (0mg THC/CBD). Drug is administered and smoked immediately prior to exposure therapy sessions 3-6. 70 participants will be randomly assigned to each treatment arm. All participants will receive prolonged exposure therapy.
  Interventions: Drug: Delta-9-tetrahydrocannabinol (THC) only
- THC:CBD 1:1 (Experimental): In a double-blind, placebo and active-controlled, between-subjects design, the investigators will administer drugs containing THC (2.5mg), CBD (2.5mg) or PBO (0mg THC/CBD). Drug is administered and smoked immediately prior to exposure therapy sessions 3-6. 70 participants will be randomly assigned to each treatment arm. All participants will receive prolonged exposure therapy.
  Interventions: Drug: THC:CBD 1:1

INTERVENTIONS:
Drug: Cannabidiol (CBD) only — Cannabis consisting of 2.5mg CBD and 0mg Delta-9-tetrahydrocannabinol (THC) is administered via smoking.
  Other Names: Cannabis
  Arms: Cannabidiol (CBD) only
Drug: Placebo only — Placebo is administered via smoking in the same way as active drugs. Placebo cannabis material obtained through National Institute of Drug Abuse (NIDA) contains 0mg THC and 0mg CBD
  Other Names: Sugar Pill
  Arms: Placebo (PBO) only
Drug: Delta-9-tetrahydrocannabinol (THC) only — Cannabis containing 2.5mg THC and 0mg CBD is administered via smoking.
  Other Names: Cannabis
  Arms: Delta-9-tetrahydrocannabinol (THC) only
Drug: THC:CBD 1:1 — Cannabis containing 2.5mg of THC and 2.5mg of CBD is administered via smoking.
  Other Names: Cannabis
  Arms: THC:CBD 1:1

SUMMARY:
The overall strategy is to recruit veterans with PTSD who report minimal current cannabis use but are interested in or considering therapeutic cannabis to manage mental health symptoms (anxiety, depression, PTSD and/or suicidality). The information gained from this study could lead to the development of new treatments for persons who suffer from post-traumatic stress disorder and maintain better mental health.

DETAILED DESCRIPTION:
The total time commitment estimated per participant 20 study visits. This is broken down below:

Visit 1: Pre-Screening and informed Consent: During this visit the potential participant will learn about the study procedures and sign the informed consent documents. Also, during this visit a licensed clinician will administer the (CAPS-5).

Visit 2: Physical Examination and Questionnaires: During this visit the participant will undergo a full physical examination conducted by a licensed medical professional. At this time, they will collect blood, urine, breathalyzer and saliva samples.

Visit 3: Baseline Assessments & Pre-Treatment Behavioral Tasks and Neurocognitive Assessments: During this visit, we will administer a baseline assessment first, then we will administer behavioral tasks that measure reward decision-making. Pre-Treatment Fear Acquisition & Extinction Learning and Magnetic Resonance (MR) Scan: During this visit the participant will complete several computer tasks, and the study staff will be measuring reaction time and psychophysiological measures. The tasks that the participant will perform will show three different images and an aversive stimulus (e.g. which will be a mild electric shock to the ankle paired with a snake hissing sound of an animated snake) may follow one image most of the time, while the other images may never be followed by the aversive cue. The participant will need to try to predict whether the aversive cue will occur or not based on which image is shown and will be asked to repeatedly rate on a scale how likely it is that he or she thinks an aversive cue will occur after each image. Lastly, during the session the participant will also be asked to report his or her level of anxiety on a scale from 0 to 100.

Visit 4: Pre-Treatment Fear Extinction Recall with MR Scan: This visit will be very similar to Visit 4. Participants will participate in the same type of task inside the MR scanner, while the study staff measures reaction time and psychophysiological responding and brain activation. Participants will view the same images he or she did previously and may experience the same aversive stimulus as during Visit 3. Participants will again be asked to rate how much they expect to experience the aversive stimulus after each image and will also be asked to report their level of anxiety on a scale from 0 to 100.

Visit 5&6: Prolonged Exposure (PE) Sessions 1 & 2: These sessions will consist of psychoeducation that includes discussion or reactions to trauma, treatment rationale, breathing retraining, and review of the Subjective Units of Distress Scale (SUDS) to assess level of distress from 0 to 100 (100=extreme anxiety/distress) when facing fears. One session occurs weekly across 2 weeks.

Visit 7-10: These sessions will consist of repeated exposures to trauma memories (imaginal exposure) and avoided situations (in vivo exposure). As is standard, patients will also practice exposures (e.g., listen to tapes of imaginal exposure, carry out in vivo exposure) outside of PE sessions as "homework". At exposure-focused sessions (Sessions 3-6) either cannabis or placebo (PBO) will be administered just before the session. One session occurs weekly across 8 weeks.

Visit 11: This visit is similar as the previous just a little longer due to a mid-treatment assessment. (Session 7)

Visit 12-14: These sessions will consist of repeated exposures to trauma memories (imaginal exposure) and avoided situations (in vivo exposure). As is standard, patients will also practice exposures (e.g., listen to tapes of imaginal exposure, carry out in vivo exposure) outside of PE sessions as "homework". At exposure-focused sessions (Sessions 8-10) either cannabis or PBO will be administered just before the session. One session occurs weekly across 8 weeks.

Visit 15: Post-Treatment Assessments: PE Session 11 will include a review of therapeutic gains/relapse prevention/assessments.

Visit 16: Post-Treatment Behavioral Tests and MR Scan: This visit will be very similar to Visit 3. Participants will participate in the same type of task inside the MR scanner, while the study staff measures reaction time and psychophysiological responding and brain activation. Participants will view the same images he or she did previously and may experience the same aversive stimulus as during Visit 3. Participants will again be asked to rate how much they expect to experience the aversive stimulus after each image and will also be asked to report their level of anxiety on a scale from 0 to 100.

Visit 17: Post- Treatment Behavioral Tests and MR Scan: This visit will be very similar to Visit 4. Participants will participate in the same type of task inside the MR scanner, while the study staff measures reaction time and psychophysiological responding and brain activation. Participants will view the same images he or she did previously and may experience the same aversive stimulus as during Visit 5. Participants will again be asked to rate how much they expect to experience the aversive stimulus after each image and will also be asked to report their level of anxiety on a scale from 0 to 100.

Visit 18: 3-Month Follow-Up Treatment Assessment: This session is similar to Visit 15 and will include review of therapeutic gains/relapse prevention/assessments.

Visit 19: 6-Month Follow-Up Treatment Assessment: This session is similar to Visit 18 and will include review of therapeutic gains/relapse prevention/assessments.

Visit 20: 9-Month Follow-Up Treatment Assessment: This session is similar to Visit 19 and will include review of therapeutic gains/relapse prevention/assessments.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to consent to the study
* Agree to comply with requirements and procedures
* Veteran who has served in a branch of the US armed forces
* Between ages 18-60
* Report using cannabis within the past three years but not more than twice in the past month
* Exposure to Criterion A stressor defined by CAPS-5 and identified by Life Events Checklist-5 (LEC-5); trauma does not have to be related to combat or military service
* Significant PTSD severity as indicated by CAPS-5 diagnosis and/or score >= 25 of at least one month prior to study entry, PTSD is patient's primary concern
* not currently receiving any psychotherapy for PTSD

Exclusion Criteria:

* Pregnant, lactating or are a heterosexually active, pre-menopausal woman who is NOT using medically approved birth control (e.g., oral or depot contraception, contraceptive implant, IUD, condom/foam, sterilization, tubal ligation)
* Current or past diagnosis of any bipolar or related disorder or schizophrenia spectrum and other psychotic disorder as determined by the SCID-5 or previous diagnosis by a licensed psychologist or psychiatrist
* Determined to be at high risk for suicide requiring immediate intervention based on the C-SSRS and/or clinician judgment
* Meet criteria for substance use disorder other than Cannabis Use Disorder or Alcohol (Mild or Moderate) or Nicotine Use Disorder, determined by the SCID-5
* Presence of contraindications, current or past allergic or adverse reaction, or known sensitivity to smoking cannabis
* Concomitant treatment with medication taken daily that has level 1 evidence indicating severe drug-drug interactions with cannabis
* Currently receiving psychotherapy for PTSD or previously received exposure-based PTSD treatment
* Current diagnosis or evidence of significant or uncontrolled hematological, endocrine, cerebrovascular, cardiovascular, systemic, pulmonary, pulmonary fibrosis, or other forms of restrictive lung disease, immunocompromising, or neurological disease
* Current diagnosis of a mood, anxiety, or other disorder that is more clinically salient than PTSD
* Cognitive exhibit impairment
* Lack of fluency in English
* Insufficient memory of the index traumatic event
* Pervasive development disorder history
* Seeking or currently undergoing treatment for Cannabis Use Disorder.
* Traumatic brain injury (TBI) with current cognitive impairment related to TBI
* Exclusively left-handed (score of -100 on Handedness Questionnaire)
* claustrophobic
* MRI contraindications (e.g., ferrous metal in head/body)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2031-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Treatment Response | Through study completion, an average of 12 months
  Clinician Administered PTSD Scale for DSM-5 (CAPS-5 Score), anxiety, mood, suicidality, disability.
  The CAPS-5 is a clinician interview that determines the presence and severity of PTSD consistent with the Diagnostic & Statistical Manual 5 (DSM-5) and allows for assessing changes in symptom severity over time. PTSD diagnosis is based on meeting the DSM-5 symptom cluster criteria (minimum threshold of symptoms with a score ≥ 2) with a qualifying criterion A index trauma. The CAPS-5 Total Severity Score is calculated by summing the total score for each of the four symptom categories to assess past-month PTSD symptoms on a specific traumatic event: intrusion (Category B), Avoidance (Category C), Mood and Cognition (Category D), and Hyperarousal (Category E). CAPS-5 Total Severity scores range from 0-80, where higher scores indicate worse PTSD severity.

SECONDARY OUTCOMES:
Brain measures | Pre and post treatment-Through study completion, an average of 12 months
  Functional magnetic resonance imaging (fMRI) will be used to measure blood oxygen level dependent (BOLD) changes in regions of interest (amygdala, ventromedial prefrontal cortex, hippocampus) during tasks.
Heart rate | through study completion, an average of 12 months
  Heart rate is taken prior to the start of prolonged exposure therapy sessions, in the middle of the session before exposure and at the end of the session.
Blood pressure | through study completion, an average of 12 months
  systolic and diastolic will be assessed before, during and after prolonged exposure therapy session. Specifically this measure is taken during drug sessions to measure the changes in physiological arousal during drug consumption.
Skin conductance response | through study completion, an average of 12 months
  Skin conductance is a measure of physiological arousal, it can be used to measure periods of heightened emotional responses to stimuli, here it is used to confirm fear conditioning.
Drug Effects Questionnaire (DEQ) | through study completion, an average of 12 months
  Subjective ratings of drug effects on from 1-5 on the following scale: "feel", "high", and "like"
Visual Analogue Scale of Mood (VAS) | through study completion, an average of 12 months
  Subjective ratings of mood and drug effects on a 0-100 scale. Higher numbers on the scale reflect stronger experiences of different mood and drug effects. Each item is scored individually. There is no overall score.
Quality of Life Inventory (QOLI) | through study completion, an average of 12 months
  assessment of well-being and satisfaction of life. The questionnaire is a 32-item scale ranging from -6 (extreme dissatisfaction) to +6 (extreme satisfaction). Scores range from 1-77 with higher scores indicating higher life satisfaction.
Pittsburgh Sleep Quality Index (PSQI) | through study completion, an average of 12 months
  Used to evaluate overall sleep quality. Participants rate sleep quality on a 4 point scale from 0 - "not during the last month" to 3 - "three or more times per week" relating to various sleep concerns. Scores range from 1-21 with higher scores indicating worse sleep quality.
Epworth Sleepiness Scale (ESS) | through study completion, an average of 12 months
  assessment of daytime sleepiness in adults. Participants rate feeling sleepy during various activities on a 4 point scale from 0 - "no chance of dozing" to 3 - "high chance of dozing". Scores range from 0-24 and are characterised as follows: 0-7:It is unlikely that you are abnormally sleepy. 8-9:You have an average amount of daytime sleepiness. 10-15:You may be excessively sleepy depending on the situation. You may want to consider seeking medical attention.
  16-24:You are excessively sleepy and should consider seeking medical attention.
Brief Pain Inventory (BPI) | through study completion, an average of 12 months
  assessment of the severity of pain and its impact on functioning. The scale consists of nine questions with a mixture of visual analogue scales and written answers. Questions 3-6 measure current pain levels on a scale from 1 - "no pain" to 10 "pain as bad as you can imagine" with higher ratings suggesting greater levels of pain (range 0-40). Question 9 has 7 nested questions (rated from 0 - 'Does not interfere" to 10 - "Completely interferes") relating to how much pain is interfering with mood, everyday tasks and sociability (range 0-70), a higher rating indicates greater issues arising from pain.
Short form 36 | through study completion, an average of 12 months
  assessment of general health questions. Each question is scored on a range from 0-100 with higher scores indicating a more favourable health state.
fMRI | through study completion, an average of 12 months
  using fMRI we can look at the differences between individuals during fear processing responses.
Psychophysiology | through study completion, an average of 12 months
  Skin conductance response (SCR): change in SCR [peak amplitude from 0.5-4.5 sec following stimulus presentation minus average 2 second baseline prior to stimulus presentation].
DNA analysis | through study completion, an average of 12 months
  Plasma samples collected are analyzed for genetic and epigenetic markers of endocannabinoid system functioning.
Cannabinoid concentration - Blood | through study completion, an average of 12 months
  As well as measuring drug levels during treatment, blood samples allow us to track the activity of the endocannabinoid system throughout the treatment. A novel approach to determine whether Delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD) function differently in the endocannabinoid system.
Drug/Pregnancy tests | through study completion, an average of 12 months
  Urine samples are also provided on regular visits for drug testing and pregnancy testing.
Cannabinoid concentration - Salvia | through study completion, an average of 12 months
  As well as measuring drug levels during treatment, these samples allow us to track the activity of the endocannabinoid system throughout the treatment. A novel approach to determine whether Delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD) function differently in the endocannabinoid system.

CONTACTS AND LOCATIONS:
Locations (1):
- Tolan Park Medical Building, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided